CLINICAL TRIAL: NCT05265897
Title: Improving Implementation of Lung Cancer Screening in Diverse Populations II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Kristina Anne Crothers, Professor, SOM: Department of Medicine: Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SITE00000215
Record Dates: First submitted 2022-02-04; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Early Detection of Cancer; Lung Cancer
Keywords: lung cancer screening; low-dose chest CT scan
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Alternating intervention controlled trial where treatment assignment was alternated weekly.
  Participants who underwent baseline or annual lung cancer screening were assigned to receive a mailing within one week of their scan, either: 1) usual care: a brief form letter with screening results; or 2) usual care plus "Commonly Asked Questions" informational document (intervention).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Brief form letter with lung cancer screening results
- CAQ (Experimental): Usual care, plus "Commonly Asked Questions after Lung Cancer Screening" informational document (CAQ)
  Interventions: Other: CAQ

INTERVENTIONS:
Other: CAQ — Informational document
  Arms: CAQ

SUMMARY:
This project assesses the feasibility, appropriateness, and acceptability of a "Commonly Asked Questions after Lung Cancer Screening" (CAQ) informational document that the investigators created, resulting from patient and provider discussion in focus groups and interviews. If effective, the CAQ may be a new tool to help improve patient understanding of LCS results and adherence to follow-up recommendations.

DETAILED DESCRIPTION:
Barriers to optimal implementation of lung cancer screening (LCS) include low levels of patient knowledge. Patient understanding of LCS results may alleviate distress and improve understanding of recommendations. The investigators developed a "Commonly Asked Questions after LCS" (CAQ) information sheet based on gaps in knowledge identified by patient focus groups and provider interviews. The study objective was to assess CAQ appropriateness and acceptability, and preliminary impact on patient understanding and distress after receiving LCS results.

The investigators conducted a pilot alternating intervention controlled trial of the CAQ. All patients in the University of Washington/Seattle Cancer Care Alliance LCS program who underwent baseline or annual LCS were received a mailing within one week of their scan, either: 1) usual care: a brief form letter with screening results; or 2) usual care plus the CAQ (intervention). The mailing assignment was alternated weekly. Mailed follow-up surveys assessed appropriateness and acceptability of CAQ as well as LCS knowledge in the intervention group.

Primary outcomes include: 1) Ratings of "I understand the results of my most recent LCS CT scan" on a Likert Scale; 2) Correct self-report of next step based on Lung-RADS standardized follow-up; 3) symptoms of distress (measured by IES); as well as 4) measures of acceptability and appropriateness. Secondary outcomes include responses to 6 questions regarding lung cancer screening knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone LCS or is referred for LCS
* Able to give informed consent

Exclusion Criteria:

* Cognitive or language limitations (i.e., expressive language limitations, non-English speaking
* Known malignancy other than non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Understanding | 1 week post-randomization
  Ratings of "I understand the results of my most recent LCS CT scan" on a Likert Scale
Patient Next Step | 1 week post-randomization
  Correct self-report of next step based on Lung-RADS standardized follow-up
Patient Distress | 1 week post-randomization
  Symptoms of distress based on Impact of Event Scale (IES)
CAQ Appropriateness and Acceptability | 1 week post-randomization
  Survey questions soliciting patient opinion of CAQ

SECONDARY OUTCOMES:
Other Patient Knowledge and Understanding | 1 week post-randomization
  Survey questions regarding knowledge and understanding of essential components of lung cancer screening and results

CONTACTS AND LOCATIONS:
Overall Officials: Kristina A Cothers, MD, Principal Investigator — University of Washington
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

REFERENCES:
- [Derived] Triplette M, Kross EK, Snidarich M, Shahrir S, Hippe DS, Crothers K. An alternating-intervention pilot trial on the impact of an informational handout on patient-reported outcomes and follow-up after lung cancer screening. PLoS One. 2024 Apr 10;19(4):e0300352. doi: 10.1371/journal.pone.0300352. eCollection 2024. PMID 38598511